CLINICAL TRIAL: NCT05328947
Title: Normative Biomechanical Measures of Reaching in Able-Bodied Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Kristin Zhao, PhD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 22-000958
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Individuals With Functional Limitations Which May Impact Their Forward Reach

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normal Controls (Experimental)
  Interventions: Other: Modified Functional Reach and Functional Reach

INTERVENTIONS:
Other: Modified Functional Reach and Functional Reach — Establishment of Modified Functional Reach Test (mFRT) and Function Reach Test (FRT) values for individuals with no functional impairments.

SUMMARY:
A study to obtain normative values and repeatability measures during functional reaching tasks in able-bodied individuals with no functional limitations.

DETAILED DESCRIPTION:
The study has three main aims: 1) Define the data collection methods, and calculate the repeatability, of joint angles, muscle activation magnitudes, seating pressure, foot pressure, and reach distance during seated and standing reaching activities. 2) Collect normative values of joint angles, muscle activation magnitudes, seating pressure, foot pressure, and reach distance during seated and standing functional reaching tasks in 40 participants with no functional limitations. Descriptive statistics will include calculating the mean, median, standard deviation, and range of the outcome variable values. 3) Compare joint angles, muscle activation magnitudes, seating pressure, foot pressure, and reach distance collected during a seated reaching task to those collected during a standing reaching task.

The data collected may be used in the future as baseline reference and repeatability values of outcome measures against which to compare values from individuals with functional limitations to quantify their functional ability.

ELIGIBILITY:
Inclusion Criteria:

• 20-59 years of age at time of enrollment

Exclusion Criteria:

* Failure to give consent or follow simple commands
* Score of 7 or above on the QuickDASH Outcome Measure
* Score of 5 or above on the Oswestry Low Back Disability Questionnaire
* Score of 76 or below on the Lower Extremity Functional Scale
* Diagnosis of a neuromuscular disorder (e.g., muscular dystrophy, multiple sclerosis, fibromyalgia)
* Diagnosis of an inner ear balance disorder (e.g., benign paroxysmal positional vertigo)
* Insufficient active range of motion of bilateral shoulders or hips that results in inability to perform forward or lateral reaching tasks
* Any illness or condition which, based on the research team's assessment, will compromise the patient's ability to comply with the protocol, patient safety, or the validity of the data collected during this study

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Joint angles | One data collection session, lasting approximately 4 hours
  Change in measurements of joint angles at the shoulders, hips, knees, and ankles, measured in degrees.
Electromyography | One data collection session, lasting approximately 4 hours
  Muscle activity over time and peak muscle activity, measured in volts. Muscles measured: erector spinae, rectus abdominis, gluteus maximus, gluteus medius, medial hamstring, vastus lateralis, gastrocnemius, and tibialis anterior.
Center of pressure excursion | One data collection session, lasting approximately 4 hours
  Path of movement of the center of pressure applied by the buttocks to the seating surface and applied by the feet to the floor.
Seated and foot pressures | One data collection session, lasting approximately 4 hours
  Plot of pressure magnitude over the surface of the buttocks and the bottom of the feet.
Reach distance | One data collection session, lasting approximately 4 hours
  Measurement of the furthest distance reached, measured in centimeters.

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No